CLINICAL TRIAL: NCT02918890
Title: Intensive Unimanual (CIMT) and Bimanual Training (HABIT) in Children With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-140
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy; Hemiplegia; Children
Keywords: Pediatric; HABIT; CIMT; Cerebral Palsy; Hemiplegia; Children; Therapy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia; Habits | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Constraint Induced Movement Therapy (Experimental): Procedure: Constraint-Induced Movement Therapy 90 hours Other Name: CIT, CI Therapy, restraint therapy, PT, OT, rehab
  Interventions: Other: Constraint-induced Movement Therapy
- Hand-Arm Bimanual Intensive Therapy (Experimental): Procedure: Hand-Arm Bimanual Intensive Therapy (HABIT) 90 hours Other Name: HABIT, bimanual training, bilateral training, restraint therapy, PT, OT, rehab
  Interventions: Other: Hand-arm Bimanual Intensive Therapy

INTERVENTIONS:
Other: Constraint-induced Movement Therapy
  Arms: Constraint Induced Movement Therapy
Other: Hand-arm Bimanual Intensive Therapy
  Arms: Hand-Arm Bimanual Intensive Therapy

SUMMARY:
A randomized control trial examining the relationship between changes in hand function and brain plasticity following intensive therapy. Two treatment approaches are used: constraint-induced movement therapy (CIMT) or Hand-Arm Bimanual Intensive Therapy (HABIT). The protocols have been developed at TC Columbia University to be child friendly and draw upon our extensive experience with constraint-induced movement therapy in children with cerebral palsy. Our center has been providing interventions camps for children with cerebral palsy since 1998. The interventions are performed in a 15 day day-camp setting with several children and at least one interventionist per child. The aim of the intervention is to improve the use of the affected hand and quality of overall movement in a fun, social setting. PARTICIPATION IS FREE. Please check out our website for more information: http://www.tc.edu/centers/cit/

DETAILED DESCRIPTION:
Constraint-induced Movement Therapy and Bimanual training are motor-learning based approaches to engage children in fun activities. This study looks at what areas of the brain are responsible for recovery after intensive training. We are trying to understand how the brain responds to movement training and hope that in the future we can develop new treatments for hemiplegia based on what we learn about the brain in this study.

To study the areas of the brain we will use Magnetic Resonance Imaging (MRI) to take pictures of the brain and Transcranial Magnetic Stimulation (TMS) to determine parts of the brain involved in using the hand. TMS uses a brief magnetic field over the scalp by using a wand that looks like a figure 8. The wand can make brief magnetic fields over a series of spots on your child's head to activate the brain cells under the wand. Non-invasive, single pulse TMS will be used in this study, which is considered minimal risk and tolerable to children. If your child has a recurrent history of seizures after two years of age, he/she might not qualify.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral cerebral palsy

Exclusion Criteria:

* Current medical illness unrelated to CP
* Seizure disorder
* Current use of medications know to lower the seizure threshold
* Metallic object(s) in body, other than dental fillings
* Pregnancy
* Claustrophobia

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gordon, Ph.D., Principal Investigator — Teachers College, Columbia University; Kathleen Friel, Ph.D., Principal Investigator — Burke Neurological Institute
Locations (1):
- Teachers College, Columbia University Center for Cerebral Palsy Research, New York, New York, United States

REFERENCES:
- [Background] Charles J, Gordon AM. Development of hand-arm bimanual intensive training (HABIT) for improving bimanual coordination in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2006 Nov;48(11):931-6. doi: 10.1017/S0012162206002039. PMID 17044964
- [Background] Gordon AM. To constrain or not to constrain, and other stories of intensive upper extremity training for children with unilateral cerebral palsy. Dev Med Child Neurol. 2011 Sep;53 Suppl 4:56-61. doi: 10.1111/j.1469-8749.2011.04066.x. PMID 21950396
- [Result] Charles JR, Wolf SL, Schneider JA, Gordon AM. Efficacy of a child-friendly form of constraint-induced movement therapy in hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2006 Aug;48(8):635-42. doi: 10.1017/S0012162206001356. PMID 16836774
- [Result] Gordon AM, Charles J, Wolf SL. Efficacy of constraint-induced movement therapy on involved upper-extremity use in children with hemiplegic cerebral palsy is not age-dependent. Pediatrics. 2006 Mar;117(3):e363-73. doi: 10.1542/peds.2005-1009. PMID 16510616
- [Result] Gordon AM, Schneider JA, Chinnan A, Charles JR. Efficacy of a hand-arm bimanual intensive therapy (HABIT) in children with hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2007 Nov;49(11):830-8. doi: 10.1111/j.1469-8749.2007.00830.x. PMID 17979861
- [Result] Gordon AM, Hung YC, Brandao M, Ferre CL, Kuo HC, Friel K, Petra E, Chinnan A, Charles JR. Bimanual training and constraint-induced movement therapy in children with hemiplegic cerebral palsy: a randomized trial. Neurorehabil Neural Repair. 2011 Oct;25(8):692-702. doi: 10.1177/1545968311402508. Epub 2011 Jun 23. PMID 21700924
- [Result] Friel KM, Ferre CL, Brandao M, Kuo HC, Chin K, Hung YC, Robert MT, Flamand VH, Smorenburg A, Bleyenheuft Y, Carmel JB, Campos T, Gordon AM. Improvements in Upper Extremity Function Following Intensive Training Are Independent of Corticospinal Tract Organization in Children With Unilateral Spastic Cerebral Palsy: A Clinical Randomized Trial. Front Neurol. 2021 May 3;12:660780. doi: 10.3389/fneur.2021.660780. eCollection 2021. PMID 34012418

RESULTS

PARTICIPANT FLOW:
Groups:
- CIMT: Procedure: Constraint-Induced Movement Therapy 90 hours Other Name: CIT, CI Therapy, restraint therapy, PT, OT, rehab
  Constraint-induced Movement Therapy
- HABIT: Procedure: Hand-Arm Bimanual Intensive Therapy (HABIT) 90 hours Other Name: HABIT, bimanual training, bilateral training, restraint therapy, PT, OT, rehab
  Hand-arm Bimanual Intensive Therapy
Period: Overall Study
Arm/Group | CIMT | HABIT
Started | 41 | 42
Contralateral | 7 | 3
Ipsilateral | 26 | 30
Bilateral | 7 | 6
Completed | 41 (We were unable to complete TMS or DTI on 1 participant so only data for 40 participants with CST determination were included.) | 41 (We were unable to complete TMS or DTI on 2 participants so only data for 39 participants with CST determination were included.)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant (CIMT) and 2 participants (HABIT) were excluded from analysis due to inability to determine corticospinal tract laterality
Groups:
- Total: Total of all reporting groups
Arm/Group | CIMT | HABIT | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.33 (2.83) | 9.58 (3.42) | 9.46 (3.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 27 | 21 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 37 | 37 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 26 | 30 | 56
  More than one race | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Jebsen-Taylor Test of Hand Function [Mean (Standard Deviation); unit: seconds] — The JTTHF measures the time taken to complete six unimanual tasks, which include flipping cards, moving small objects, and lifting cans. The total score is the amount of time taken to complete all tasks. The test was performed on both the more affected and less affected hands. The JTTHF is well-validated and has excellent reliability.
  seconds | 405.1 (306.8) | 402.5 (296.5) | 403.8 (299.85)
Assisting Hand Assessment [Mean (Standard Deviation); unit: logits] — The AHA is a validated test for measuring bimanual hand use in children with upper extremity impairments. The AHA measures the use of the more affected hand in bimanual activities during a play-like testing session. Sessions were videotaped and scored off-site by a blinded evaluator. The AHA has excellent validity, reliability (0.97-0.99) and responsiveness to change. The AHA units were used for the analysis. The smallest detectable difference (SDD) for AHA is an improvement of at least 5 units.
  logits | 56.7 (20.7) | 55.2 (8.7) | 56.0 (15.83)
Box and Blocks Test [Mean (Standard Deviation); unit: blocks] — The BBT measures how many blocks (2.5 cm3) an individual can move from one box, over a barrier, to an adjacent box in one minute. Both hands were tested. The BBT is valid and reliable for children with CP.
  blocks | 18.2 (10.1) | 16.6 (9.8) | 17.4 (9.94)
Canadian Occupational Performance Measure - Performance [Mean (Standard Deviation); unit: units on a scale] — The COPM is a structured interview in which the individuals are asked to identify up to five functional goals. In this study, parents reported their child's functional goals. Parents rated how well children perform each goal (COPM-Performance), and how satisfied they were with the child's performance (COPM-Satisfaction). The same caregiver was interviewed before and after the intervention. A change of 2 or more points in each scale of COPM is considered a minimum clinically important difference (MCID). The COPM has been validated for parents of children with disabilities.
  units on a scale | 2.9 (1.1) | 3.0 (1.4) | 2.95 (1.07)
Canadian Occupational Performance Measure - Satisfaction [Mean (Standard Deviation); unit: units on a scale] — The COPM is a structured interview in which the individuals are asked to identify up to five functional goals. In this study, parents reported their child's functional goals. Parents rated how well children perform each goal (COPM-Performance), and how satisfied they were with the child's performance (COPM-Satisfaction). The same caregiver was interviewed before and after the intervention. A change of 2 or more points in each scale of COPM is considered a minimum clinically important difference (MCID). The COPM has been validated for parents of children with disabilities.
  units on a scale | 3.1 (1.6) | 3.3 (1.8) | 3.2 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Jebsen-Taylor Test of Hand Function
Description: The JTTHF measures the time taken to complete six unimanual tasks, which include flipping cards, moving small objects, and lifting cans. The total score is the amount of time taken (in seconds) to complete all tasks. A lower score means a better outcome.
Time Frame: Baseline (pre-test), within 2 days after treatment (post-test), 6 months after treatment (follow-up)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- CIMT; Contralateral CST: Constraint Induced Movement Therapy; contralateral corticospinal tract
- CIMT; Ipsilateral CST: Constraint Induced Movement Therapy; ipsilateral corticospinal tract
- CIMT; Bilateral CST: Constraint Induced Movement Therapy; bilateral corticospinal tract
- HABIT; Contralateral CST: Hand Arm Bimanual Intensive Training; contralateral corticospinal tract
- HABIT; Ipsilateral CST: Hand Arm Bimanual Intensive Training; ipsilateral corticospinal tract
- HABIT; Bilateral CST: Hand Arm Bimanual Intensive Training; bilateral corticospinal tract
Arm/Group | CIMT; Contralateral CST | CIMT; Ipsilateral CST | CIMT; Bilateral CST | HABIT; Contralateral CST | HABIT; Ipsilateral CST | HABIT; Bilateral CST
Number analyzed (Participants) | 7 | 26 | 7 | 3 | 30 | 6
seconds
  Pre-test; more affected hand | 323.6 [89.9 to 557.3] | 479.5 [358.5 to 600.5] | 265.6 [46.6 to 484.6] | 121.3 [-183.9 to 426.5] | 435.7 [331.2 to 540.2] | 377.3 [122.4 to 632.1]
  Post-test; more affected hand | 224 [47.4 to 400.7] | 354.1 [254.5 to 453.7] | 175.9 [-28.8 to 380.7] | 98.9 [-170.5 to 368.4] | 378.6 [281.3 to 476] | 316.8 [90.8 to 542.8]
  6 month follow-up; more affected hand | 266.1 [109.5 to 422.7] | 342.4 [233 to 451.9] | 213.3 [13.6 to 413] | 146 [-152 to 444] | 380.2 [274.2 to 486.2] | 323.8 [152 to 495.5]

2. Primary Outcome: Assisting Hand Assessment
Description: The AHA is a validated test for measuring bimanual hand use in children with UE impairments. The AHA measures the use of the more affected hand in bimanual activities during a play-like testing session. Sessions were videotaped and scored off-site by a blinded evaluator. The AHA has excellent validity, reliability (0.97-0.99) and responsiveness to change. The AHA units were used for the analysis (range 0-100). The smallest detectable difference (SDD) for AHA is an improvement of at least 5 units. A higher score means a better outcome.
Time Frame: Baseline (pre-test), within 2 days after treatment (post-test), 6 months after treatment (follow-up)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CIMT; Contralateral CST | CIMT; Ipsilateral CST | CIMT; Bilateral CST | HABIT; Contralateral CST | HABIT; Ipsilateral CST | HABIT; Bilateral CST
Number analyzed (Participants) | 7 | 26 | 7 | 3 | 30 | 6
units on a scale
  Pre-test | 55.4 [50.4 to 60.5] | 52.5 [48.5 to 56.6] | 62.3 [57.1 to 67.5] | 61.3 [57.9 to 64.8] | 54.8 [51.4 to 58.1] | 54.5 [48.1 to 60.9]
  Post-test | 58.6 [52.6 to 64.5] | 54 [50.2 to 57.8] | 63.7 [57.6 to 69.8] | 65 [57.9 to 72.1] | 57.2 [54.1 to 60.3] | 56.6 [49.4 to 63.6]
  6 month follow-up | 58.1 [52.4 to 63.9] | 54.4 [50.3 to 58.4] | 64.1 [57.8 to 70.5] | 66.3 [62.9 to 69.8] | 56.5 [53.4 to 59.5] | 56.7 [50.5 to 62.8]

3. Primary Outcome: Box and Blocks Test
Description: The BBT measures how many blocks (2.5 cm3) an individual can move from one box, over a barrier, to an adjacent box in 1 min. Both hands were tested. The BBT is valid and reliable for children with CP. A higher score means a better outcome.
Time Frame: Baseline (pre-test), within 2 days after treatment (post-test), 6 months after treatment (follow-up)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: blocks moved in 1 minute
Arm/Group | CIMT; Contralateral CST | CIMT; Ipsilateral CST | CIMT; Bilateral CST | HABIT; Contralateral CST | HABIT; Ipsilateral CST | HABIT; Bilateral CST
Number analyzed (Participants) | 7 | 26 | 7 | 3 | 30 | 6
blocks moved in 1 minute
  Pre-test; more affected hand | 18.9 [14.7 to 23.1] | 16.6 [12.1 to 21.1] | 21.4 [15 to 27.9] | 26 [19.2 to 32.8] | 16.2 [12.5 to 19.9] | 14 [7.9 to 20.1]
  Post-test; more affected hand | 25.6 [21 to 30.1] | 19.2 [13.9 to 24.4] | 27 [20.5 to 33.5] | 27 [20.6 to 33.4] | 19.2 [15.6 to 22.8] | 18.7 [10 to 27.4]
  6 month follow-up; more affected hand | 23.4 [18.7 to 28] | 19.7 [14.6 to 24.8] | 24.7 [17.4 to 31.9] | 31.3 [19.7 to 42.9] | 19.3 [15.6 to 23] | 18.2 [9.5 to 26.9]

4. Secondary Outcome: Canadian Occupational Performance Measure
Description: The COPM is a structured interview in which the individuals are asked to identify up to five functional goals. In this study, parents reported their child's functional goals. Parents rated how well children perform each goal (COPM-Performance), and how satisfied they were with the child's performance (COPM-Satisfaction). The same caregiver was interviewed before and after the intervention. A change of 2 or more points in each scale of COPM is considered a minimum clinically important difference (MCID). The COPM has been validated for parents of children with disabilities. A high score means a better outcome (range 0-10).
Time Frame: Baseline (pre-test), within 2 days after treatment (post-test), 6 months after treatment (follow-up)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CIMT; Contralateral CST | CIMT; Ipsilateral CST | CIMT; Bilateral CST | HABIT; Contralateral CST | HABIT; Ipsilateral CST | HABIT; Bilateral CST
Number analyzed (Participants) | 7 | 26 | 7 | 3 | 30 | 6
score on a scale
  Pre-Test; Performance | 2.5 [1.2 to 3.8] | 2.9 [2.5 to 3.3] | 3.2 [2.5 to 3.9] | 3.5 [3.2 to 3.7] | 2.8 [2.3 to 3.4] | 3.6 [2.9 to 4.2]
  Post-Test; Performance | 4.8 [3.3 to 6.4] | 5.7 [5 to 6.4] | 6.3 [5.3 to 7.4] | 5.9 [4.6 to 7.1] | 6.4 [5.8 to 7] | 6.5 [5 to 8.1]
  6 month follow-up; Performance | 5.3 [4.6 to 6.1] | 6 [5.3 to 6.7] | 6.6 [5.7 to 7.4] | 6.9 [5.5 to 8.4] | 6.1 [5.5 to 6.6] | 6.5 [4.9 to 8]
  Pre-Test; Satisfaction | 2.9 [1.9 to 4] | 3.2 [2.6 to 3.8] | 3 [1.8 to 4.3] | 4.4 [2.1 to 6.7] | 3.3 [2.6 to 4] | 2.7 [2.1 to 3.3]
  Post-Test; Satisfaction | 5.7 [3.8 to 7.7] | 6.4 [5.5 to 7.3] | 7.2 [6 to 8.4] | 6.1 [3.7 to 8.5] | 7 [6.4 to 7.7] | 6.8 [5.5 to 8.1]
  6 month follow-up; Satisfaction | 6.3 [5 to 7.5] | 6.6 [5.9 to 7.3] | 7.3 [6.5 to 8.2] | 7.7 [5.9 to 9.5] | 6.5 [5.8 to 7.1] | 6.8 [5.5 to 8.1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CIMT | HABIT
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 1/41 | 4/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CIMT (N=41) | HABIT (N=42)
Seizure (Nervous system disorders) | 1 | 2
Fall causing broken bone (Musculoskeletal and connective tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
There were not an equal number of participants with each CST connectivity pattern. Although we did have a large number of participants with ipsilateral connectivity, we had a small number of children with purely a contralateral pattern. However, the responsiveness of these individuals across studies is not in doubt, and the findings held true even when the contralateral and bilateral groups were combined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT02918890/Prot_SAP_000.pdf